CLINICAL TRIAL: NCT04397705
Title: Remote Monitoring of Cancer Patients Presenting With Symptoms Suggestive of Covid-19 - Pilot Phase.
Brief Title: Remote Monitoring of Cancer Patients With Suspected Covid-19
Acronym: RECAP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CFTSp186
Record Dates: First submitted 2020-05-20; First posted 2020-05-21 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: COVID; Oncology; Haematological Malignancy
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm open label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ambulatory monitoring (Experimental): Participants will be asked to wear the sensors (heart rate, respiratory rate, temperature, and pulse oximetry) for three weeks. Data will be collected from the devices but will only be reviewed retrospectively and will not be used to alter participants care.
  Interventions: Device: Patient Status Engine

INTERVENTIONS:
Device: Patient Status Engine — Wearable sensors

SUMMARY:
Since emerging in December 2019, coronavirus disease 2019 (Covid-19) has developed into an unprecedented global pandemic. The causative pathogen, the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has the potential to cause a wide range of clinical syndromes, from fever, dyspnoea and cough to respiratory failure and cardiac injury necessitating critical care support. A number of patients have a more indolent clinical course and can be safely managed in the community.

Characterising the clinical course of Covid-19 infection in the oncology population and distinguishing this from other acute oncology presentations which can mimic Covid-19 is a key unmet research need. Current standard of care for monitoring patients at high risk of chemotherapy associated neutropenic sepsis involves asking them to contact their cancer centre when they feel unwell or develop a fever. No standard of care for monitoring ambulatory Covid-19 patients has yet been established. We hypothesise that using wearable biosensors to detect patients who exhibit 'red flags' for sepsis or deterioration due to Covid-19 may allow earlier assessment and intervention. There is no current evidence for wearable biosensors in ambulatory patients receiving chemotherapy, and there is no existing research into this proposed use of biosensors in patients with suspected or confirmed Covid-19 infection.

In order to justify performing a randomised controlled study comparing standard of care with biosensor driven monitoring it is important to establish the tolerability and validity of these devices. We aim to collect patient reported outcome measures (PROMs) on tolerability and assess the reliability of data transmission to a central data collection server. We will also perform an initial analysis of physiological data and correlation with clinical events

DETAILED DESCRIPTION:
This is a pilot, single arm, open label feasibility study. This is a single centre trial based in a large tertiary cancer centre which treats patients across all solid and haematological malignancies. Patients will be recruited from all disease groups.

Patients who present with symptoms suspicious for Covid-19 who the admitting clinicians deems appropriate for outpatient management will be considered for this study.

Patients who are enrolled will undergo continuous physiological monitoring for up to three weeks. This includes continuous monitoring of heart rate, respiratory rate, temperature, activity levels (by accelerometer measurement) and twice daily pulse oximetry. The physiological data will not be reviewed in real time by clinicians and therefore will not be used to alter patients' standard care. The pulse oximetry data will be visible to patients who will be given clear guidelines to follow with regards to contacting the cancer centre hotline should values deviate from baseline.

In the pilot phase of RECAP 10-30 patients will each be monitored for up to 3 weeks and the following endpoints will be addressed:

Physiological trends and interactions predictive of clinical deterioration due to COVID-19 (Co-primary endpoint) Reliability of biosensor data collection/transmission using digital technology from patients self-isolating at home (Co-primary endpoint) Acceptability and tolerability of wearable biosensors and continuous monitoring If the pilot phase is successful we will move to a phase II study in a larger number of patients where the objective will be to refine a physiological signature predictive of clinical deterioration in COVID-19 patients so that early hospitalisation and relevant medical interventions can be arranged.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are capable of giving informed consent
2. Male or female aged 18 or over
3. Diagnosis of any solid tumour or haematological malignancy meeting one of the following criteria:

   * Current malignant diagnosis
   * Received anti-cancer treatment within the last two years
4. Emergency presentation to hospital with symptoms consistent with Covid-19 deemed to meet the criteria for Covid-19 testing by admitting clinician.
5. Deemed by the admitting clinician to be suitable for outpatient management of suspected Covid-19.
6. Stable oxygen saturations of 95% or higher at time of emergency presentation.
7. Able to complete tolerability questionnaire.
8. Able and willing to comply with twice daily pulse oximetry monitoring as outlined in section 6 of the protocol.
9. ECOG-PS <4
10. Life expectancy of greater than three months as assessed by screening investigator from review of electronic patient record.

Exclusion Criteria:

1. Patients hospitalized for more than 24 hours at initial presentation with symptoms consistent with Covid-19.
2. Pregnant patients.
3. Patients unable to give informed consent.
4. Presence of ulceration or pre-existing skin rash at site of device application (left precordium and axillae). If only one axilla affected this is not an exclusion criterion if patient is happy to apply temperature sensor to the other axilla.
5. Radiotherapy to the left chest wall either during or within the six months preceding the study. Plans for subsequent radiotherapy to commence after study completion are not an exclusion criterion. If only one axilla is within the planned radiotherapy field and patient is happy to apply temperature sensor to the other axilla this is not an exclusion criteria.
6. History of allergy or contact dermatitis to medical adhesives e.g sticking plasters, ECG electrodes.
7. Patients with pacemakers, implantable defibrillators or neurostimulators.
8. Patients who are currently receiving treatment as part of a clinical study or have had their end of treatment visit for another clinical study less than 30 days prior to the study enrollment visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Device Tolerability (Attrition) | Three weeks
  Percentage of patients who choose to stop wearing the devices before they have completed the study
Correlation of physiological data with clinical events | Over three weeks of patients wearing devices
  Correlation of sensor collected data with clinical episodes of infection. Sensor collected data includes heart rate, respiratory rate and temperature.

SECONDARY OUTCOMES:
Device Tolerability (Questionnaire) | Questionnaire at three weeks
  Percentage of participants who answer 'agree' or 'strongly agree' on a five point Likert scale to the statement 'I would be happy to wear the sensors again for the next three weeks'. This statement is included in the questionnaires completed after three weeks of wearing the device.
Device Tolerability (Semi-structured interviews) | One to four weeks after completion of wearing the device
  Device tolerability as assessed by semi-structured interviews.
Reliability of data transmission | Over three weeks of patients wearing devices
  Reliable data transmission to central hospital system expressed as a percentage of total data points collected out of target data points collected.

CONTACTS AND LOCATIONS:
Overall Officials: John Radford, Principal Investigator — The University of Manchester
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The physiological data represents a rich clinical data resource which has the potential to be valuable in other contexts to answer future unanticipated questions. We therefore propose storing this pseudoanonymised data in a Data Bank with a lifespan initially of five years with potential for extension if appropriate ethical approval is gained. This Data Bank could then be used, under ethical approval for other research in order to maximise the potential utility of the data.